CLINICAL TRIAL: NCT06718959
Title: Efficacy and Safety Evaluation of Jet Floss EX
Brief Title: Efficacy and Safety Evaluation of Jet Floss EX After 8-week Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang Dong Bixdo Health Technology Co.,Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-287-KQ-026
Record Dates: First submitted 2024-11-26; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Bleeding on Probing; Plaque; Gingival Index
Keywords: Gingival index; Bleeding on Probing; Plaque
MeSH Terms: conditions — Plaque, Amyloid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- treatment group (Experimental): subjects continued to use distributed manual toothbrush and toothpaste every morning and evening, and add used the test product (Jet Floss EX) twice a day.
  Interventions: Device: the test product (Jet Floss EX)
- control group (Active Comparator): subjects continued to use distributed manual toothbrush and toothpaste every morning and evening, and add auxiliary product (interdental brush) twice a day.
  Interventions: Other: the control product (interdental brush)

INTERVENTIONS:
Device: the test product (Jet Floss EX) — subjects continued to use distributed manual toothbrush and toothpaste every morning and evening, and add used the test product (Jet Floss EX) twice a day. Subjects used the test product (standard sprinkler, water twice) to flush all gingival margins and adjacent spaces with 440ml of water, start with water pressure gear 1 for the first time and continued with this gear after reaching the highest level that can be asapted. If felt uncomfortable, eligible subjects can adjust it to a suitable gear. The specific installation and usage of the teeth punch refer to the product instruction.
  Arms: treatment group
Other: the control product (interdental brush) — subjects continued to use distributed manual toothbrush and toothpaste every morning and evening, and add auxiliary product (interdental brush) twice a day.
  Arms: control group

SUMMARY:
This was a single center, comparison among treatments, 8-week study of the efficacy and safety of Jet Floss EX.

Totally 72 eligible subjects were recruited in this study and randomly divided into 2 groups. During wash out phase (7 days before the study), subjects used distributed manual toothbrush and toothpaste every morning and evening to replace their own products. After that, subjects screened by dentist to ensure met the inclusion criteria. During treatment phase, for group1 (treatment group), subjects continued to use distributed manual toothbrush and toothpaste every morning and evening, and add used the test product (Jet Floss EX) twice a day. For group2 (control group), subjects continued to use distributed manual toothbrush and toothpaste every morning and evening, and add used auxiliary product (interdental brush) twice a day. During the study, any other oral care products and non-emergency oral treatment were not allowed.

Test Objective:To evaluate the efficacy and safety of test product by means of intraoral exams of BOP, PD, MGI, RMNPI, hard and soft tissues exams and selfassessment.

ELIGIBILITY:
Inclusion Criteria:

* Chinese men or women aged 18-60 years old;
* In general good health at the time of the study;
* Possess a minimum of 20 scorable teeth;
* Each quadrant has ≥4 inter tooth gaps that can be inserted by interdental brush；
* RMNPI≥0.6;
* BOP≥50%;
* MGI≥1.75;
* PD≤5 mm;
* There were no diseases that will affect the test results;
* Willing and able to participate as evidenced by signing of informed consent;
* Willing to comply with all study protocol requirements.

Exclusion Criteria:

* Intending to get pregnant, pregnant, lactating or within 6 months of delivery;
* Those who have known allergies against oral care product or have severe oral disease;
* Simultaneous participating in another oral study;
* Have any fixed facial orthodontic appliances or removable partial dentures;
* Severe presence of tartar or stain which will affect the test;
* Others whose participation in the study is determined inappropriate by the dentist.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
The improvement in BOP(Bleeding on Probing) after 8 weeks of use. | 8 weeks
  After 8 weeks of treatment, when compared with the baseline, reduction percentage in the bleeding index.
The improvement in MGI (Modified Gingival Index) after 8 weeks of use. | 8 weeks
  After 8 weeks of treatment, when compared with the baseline, reduction percentage in MGI (Modified Gingival Index).
The improvement in RMNPI (Rustogi Modification of the Navy Plaque Index) after 8 weeks of use. | 8 weeks
  After 8 weeks of treatment, when compared with the baseline, reduction percentage in RMNPI (Rustogi Modification of the Navy Plaque Index) .

SECONDARY OUTCOMES:
Compare the differences in BOP(Bleeding on Probing) between the test group and the control group after 8 weeks of uses. | 8 weeks
  Dentists evaluate the bleeding index of all study participants according to the BOP (Bleeding on Probing) evaluation criteria using CPI (Community Periodontal Index) probes. The scoring criteria are: 0= no bleeding, 1= bleeding. Calculate the percentage of sites that bleed after probing out of the total number of sites evaluated.
  The effectiveness of the water flosser(Jet Floss EX) in the test group will be analyzed by comparing the bleeding index with that of the interdental brush in the control group to determine if there are significant intergroup differences.
Compare the differences in PD (Probing Depth) between the test group and the control group after 8 weeks of uses. | 8 weeks
  Dentists evaluate the PD periodontal probing depth for all study participants. Measure the distance from the gingival margin to the bottom of the pocket on the buccal and lingual aspects at the distal, central, and mesial sites, recording six sites per tooth. Calculate the average value.
  The effectiveness of the water flosser(Jet Floss EX) in the test group will be analyzed by comparing the PD (Probing Depth) with that of the interdental brush in the control group to determine if there are significant intergroup differences.
Compare the differences in MGI (Modified Gingival Index) between the test group and the control group after 8 weeks of uses. | 8 weeks
  Dentists score the gingival condition of all study participants based on the modified gingival index criteria.
  Examine and record the MGI score on the buccal and lingual aspects at the distal, central, and mesial sites of teeth, calculate the average value.
  The effectiveness of the water flosser(Jet Floss EX) in the test group will be analyzed by comparing the PD (Probing Depth) with that of the interdental brush in the control group to determine if there are significant intergroup differences.
Compare the differences in RMNPI (Rustogi Modification of the Navy Plaque Index) between the test group and the control group after 8 weeks of uses. | 8 weeks
  Dentists evaluate the plaque condition of all study participants based on the RMNPI Modified Plaque Index using visual inspection.
  Participants should stain their teeth with a disclosing agent before evaluation.
  The teeth are divided into nine regions A-I, and plaque is scored for each region (buccal and lingual aspects of regions A-I), with the scoring criteria being: 0= no plaque; 1= plaque present. Calculate the average value.
  The effectiveness of the water flosser(Jet Floss EX) in the test group will be analyzed by comparing the PD (Probing Depth) with that of the interdental brush in the control group to determine if there are significant intergroup differences.
Evaluate the safety of the test product(Jet Floss EX) by conducting an examination and assessment of the oral soft and hard tissues after 8 weeks of uses. | 8 weeks
  Dentists will conduct an assessment of the oral soft and hard tissues for all study participants. This examination includes the inspection of the soft palate, hard palate, gingival mucosa, buccal mucosa, mucogingival fold area, tongue, sublingual and submandibular regions, salivary glands, tonsils, and the pharyngeal area.The scoring criteria are: 0= normal, 1= unnormal.
Subject satisfaction evaluation | 8 weeks
  The participants received a questionnaire at the last visit, which mainly included the improvement effect of the product.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Sino-German Union Cosmetic Institute Co., Ltd., Chaoyang District, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No